CLINICAL TRIAL: NCT00743002
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled Study of TT223 in Patients With Type 2 Diabetes Treated With Metformin and/or TZD
Brief Title: A Trial of TT223 in Patients With Type 2 Diabetes Who Are Taking Metformin and/or Thiazolidinedione
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GIN-201
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: TT223
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TT223 with Metformin and/or TZD (Experimental): TT223 as a treatment for Type 2 diabetes is administered by injection once daily at 1 mg, 2 mg and 3 mg patients currently treated with Metformin and/or Thiazolidinedione (TZD).
  Interventions: Drug: TT223 with Metformin and/or TZD
- Placebo with Metformin and/or TZD (Placebo Comparator): Placebo as a comparator is administered by injection once daily at 1 mg, 2 mg and 3 mg patients currently treated with Metformin and/or Thiazolidinedione (TZD).
  Interventions: Drug: Placebo with Metformin and/or TZD

INTERVENTIONS:
Drug: TT223 with Metformin and/or TZD — Daily subcutaneous injection: 1 mg for 1 week; followed by 2 mg for 1 week; followed by 3 mg for 10 weeks
  Arms: TT223 with Metformin and/or TZD
Drug: Placebo with Metformin and/or TZD — Daily subcutaneous injection: 1 mg for 1 week; followed by 2 mg for 1 week; followed by 3 mg for 10 weeks
  Arms: Placebo with Metformin and/or TZD

SUMMARY:
This trial is designed to show the effect of treatment with TT223 or placebo on blood glucose control after 12 weeks of treatment with a 6 month follow-up. TT223 is administered by injection once daily to patients currently treated with Metformin and/or Thiazolidinedione.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes for at least 6 months
* Treated with metformin and/or thiazolidinediones with stable dose for at least 3 months
* BMI of 21-45 kg/m2, inclusive
* HbA1c level of 7.50 - 10.00%, inclusive
* If a female of childbearing potential, willing to utilize contraception from Screening through 4 weeks after the last dose of study drug

Exclusion Criteria:

* Treatment with insulin, sulfonylurea, DPP-4 inhibitors, Symlin® and/or GLP-1 analogues ≤ 3 months prior to the Screening
* Severe hypoglycemia ≤ 60 days prior to the Screening visit or currently diagnosed with having hypoglycemia unawareness
* History of peptic ulcer(s) and/or gastrointestinal bleeding/perforation
* Previous gastric surgery, including gastric bypass, or has gastric bypass/other major surgery planned to occur during the 10 month trial
* Myocardial infarction within the last 2 years, current congestive heart failure with NYHA class 2 or greater, or chronic atrial fibrillation
* Current clinically significant and/or chronic illness
* Takes regular courses of non-steroidal anti-inflammatory drugs (NSAIDS). If these medications are discontinued upon starting Screening procedures and are not planned to be regularly used during the trial, the patient will be allowed to enter the Study
* Use of systemic corticosteroids (oral, suppository, injected). Use of inhaled or topical corticosteroids is permitted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of TT223 as a treatment for Type 2 diabetes at 1 mg, 2 mg and 3 mg. | For the duration of the trial.

SECONDARY OUTCOMES:
To evaluate the efficacy of TT223 as a treatment for Type 2 diabetes by comparing the change in HbA1c value from baseline between the TT223 and placebo groups. | For the duration of the trial.
To evaluate the efficacy of TT223 on beta cell function by assessing additional outcome measures including fasting blood glucose levels, and meal tolerance testing. | For the duration of the trial.
To determine the pharmacokinetic (PK) parameter profile of TT223 in a subset of patients. | Day 1 and Week 12 of treatment.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Artesia, California
  - Los Angeles, California
  - Santa Ana, California
  - Torrence, California
  - Walnut Creek, California
  - DeLand, Florida
  - Bloomingdale, Illinois
  - Grand Rapids, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Clifton, New Jersey
  - Asheboro, North Carolina
  - Wilmington, North Carolina
  - Bensalem, Pennsylvania
  - Athens, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Texas
  - San Antonio, Texas